CLINICAL TRIAL: NCT01093066
Title: Prospective Multicentric Evaluation of a Bladder Preservation Strategy Using a Combination of Neoadjuvant Chemotherapy and Optimal Bladder Transurethral Resection in Patients With a Urothelial Carcinoma
Brief Title: Prospective Multicentric Evaluation of a Bladder Preservation Strategy
Acronym: ReChiVe
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in the inclusion and follow-up of patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0908038; 2009-014264-19 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Urothelial Carcinoma
Keywords: urothelial carcinoma; TURB; chemotherapy
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgical resection and chemotherapy (Experimental): Maximal and optimal TURB using a standardized procedure. The TURB will always try to be optically complete.
  Neoadjuvant chemotherapy for 3 months with the intensified MVAC (6 cycles administered every 2 weeks): METHOREXATE: 30 mg/m2 D1 - VINBLASTINE: 3 mg/m2 D2 - ADRIAMYCINE 30 mg/m2 D2 - CISPLATINE 70 mg/m2 D2. + G-CSF: 5 µg/kg from D4 to D10 New maximal standardized TURB at the end of the chemotherapy. In case of a lesion localized at the bladder dome, and if a maximal TURB appears to be unsafe, a partial cystectomy without lymph node dissection will be performed.
  Interventions: Drug: optimal TURB

INTERVENTIONS:
Drug: optimal TURB — The TURB will always try to be optically complete.

SUMMARY:
Radical cystectomy is the treatment of choice for bladder infiltrative urothelium carcinoma. But the removal of the bladder reservoir has a major impact of the Quality of life. Neoadjuvant chemotherapy has been shown to be associated with an absolute 5% survival benefit. Two monocentric studies suggest that this neoadjuvant chemotherapy could be used in combination with an optimal transurethral bladder resection, in a strategy of bladder preservation, provided a complete response being obtained (about 50% in every trial using neoadjuvant MVAC protocol before a radical cystectomy). In those both studies with patients T2 to T4, the 5 years overall survival is above 65%, with more than 40% bladder preservation rate at 5 years.

The feasibility and the efficacy of such an attitude in a multicentric trail using the most active regimen (in term of complete response in metastatic patients) is unknown. The chosen regimen is therefore the intensified MVAC which allows, with the use of G-CSF, to double the dose-intensity of Adriamycin and Cisplatinum, and to decrease by 30% the methotrexate and vinblastine dose-intensity.

The efficacy and safety confirmation of such an approach could lead to consider it in patients motivated to retain a functional bladder.

DETAILED DESCRIPTION:
Every patient having signed the inform consent will have the following steps Maximal and optimal TURB using a standardized procedure. The TURB will always try to be optically complete.

Neoadjuvant chemotherapy for 3 months with the intensified MVAC (6 cycles administered every 2 weeks): METHOREXATE: 30 mg/m2 D1 - VINBLASTINE: 3 mg/m2 D2 - ADRIAMYCINE 30 mg/m2 D2 - CISPLATINE 70 mg/m2 D2. + G-CSF: 5 µg/kg from D4 to D10 New maximal standardized TURB at the end of the chemotherapy. In case of a lesion localized at the bladder dome, and if a maximal TURB appears to be unsafe, a partial cystectomy without lymph node dissection will be performed.

If a complete response is obtained (no tumor cells in the bladder muscle on the last TURB), a surveillance will be proposed without any further treatment.

Otherwise (tumor cells in the bladder muscle at the second TURB), a radical cystectomy will be done.

If the balder is spared, the follow up will be as follow: clinical examination, CT, bladder endoscopy and urinary cytology every 6 months. The possible non muscle infiltrative bladder relapses will be treated according

ELIGIBILITY:
Inclusion Criteria:

* T2 clinical stage (no palpable mass under anesthesia after TURB) Absence of diffuse Cis (Cis on random bladder biopsies) Patients above 18, and below 70 years of age PS status ≤ 2 No previous treatment for a bladder muscle infiltrative carcinoma. Previous endovesical instillations for non muscle infiltrative lesions (pTa, pT1, Cis) are allowed.

No metastases on tauraco-abdomina-pelvic CT scan (no node > 1 cm) and bone scan.

Normal biological values: neutrophils > 1,5.109 /l, platelets > 100. 109 /l, Alkaline Phosphatases < 2 x N, bilirubin < 1,5 N, Transaminases < 1,5 x N, Creatinine clearance ≥ 60 ml/min Signed inform consent Patient belonging to a social security system.

Exclusion Criteria:

All other histology than urothelial carcinoma:

* primitive adenocarcinoma
* epidermoid carcinoma
* little cells carcinoma In situ diffuse carcinoma associated with urothelial carcinoma muscular infiltrating Tumor stade > T2, T3 or T4 or pT4a (prostatitis) Serious cardiac, pulmonary, hepatitic, renal, digestive or neurological pathology which is non equilibrating or potential aggravating risk by treatment Cancer history or other actual cancer (except skin cancer) not remission or with an end of treatment inferior to 2 years Participation to another clinical trial in a delay inferior to 30 days

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2010-09-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the 5 years bladder preservation rate (with or without intravesical non muscle infiltrative recurrences, treated by TURB only or intravesical instillations of either BCG or mytomicin C). | 5 years

SECONDARY OUTCOMES:
proportion of complete response | 6 months
Chemotherapy tolerance in a neoadjuvant setting using the intensified MVAC | 3 months
Secondary cystectomy rate | 6 months
Progression free survival (either infiltrative [≥ T2] or metastatic) | 5 years
Overall bladder preservation rate | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, MD, Principal Investigator — clinique Mutualiste chirurgicale
Locations (31):
- France (31):
  - CH du Pays d'Aix-en-Provence, Aix-en-Provence
  - Clinique AXIUM - AIX EN PROVENCE, Aix-en-Provence
  - CHU Bordeaux, Bordeaux
  - Clinique Saint-Augustin, Bordeaux
  - Institut Bergonie, Bordeaux
  - CHU Caen, Caen
  - Crlcc Francois Baclesse, Caen
  - CHU Créteil, Créteil
  - Polyclinique Du Cotentin, Équeurdreville-Hainneville
  - Polyclinique de Lisieux, Lisieux
  - APHM - Marseille - Hôpital de la Conception, Marseille
  - APHM - Marseille - Hôpital la Timone, Marseille
  - CRLC Marseille, Marseille
  - Hôpital Européen - Marseille, Marseille
  - Hôpitaux privés de Metz, Metz
  - Chu Nancy, Nancy
  - Crlc Nancy, Nancy
  - Chu Nantes, Nantes
  - APHP - Saint-Louis, Paris
  - APHP- Hôpital Tenon, Paris
  - CHU Poitiers, Poitiers
  - Chu Reims, Reims
  - Institut Jean Godinot - Reims, Reims
  - Clinique Mutualiste Chirurgicale, Saint-Etienne
  - CHU Saint-Etienne, Saint-Etienne
  - ICO - SITE Gauducheau - ICL Nantes, Saint-Herblain
  - ICLN, Saint-Priest-en-Jarez
  - Hôpitaux du Léman - Thonon-les-Bains, Thonon-les-Bains
  - CHI Toulon, Toulon
  - CHU Toulouse, Toulouse
  - INSTITUT CLAUDIUS REGAUD - CRLC Toulouse, Toulouse